CLINICAL TRIAL: NCT03207750
Title: Immunogenicity, Reactogenicity and Safety Study of Pediarix®, Hiberix® and Prevenar 13® Co-administered With Two Different Formulations of GSK Biologicals' HRV Vaccine (444563) in Healthy Infants 6-12 Weeks of Age
Brief Title: This Study Will Evaluate the Immunogenicity, Reactogenicity and Safety of the Routine Infant Vaccines Pediarix®, Hiberix® and Prevenar 13® When Co-administered With GlaxoSmithKline (GSK) Biologicals' Liquid Human Rotavirus Vaccine (HRV) as Compared to GSK's Licensed Lyophilized Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201663; 2016-003210-27 (EudraCT Number)
Record Dates: First submitted 2017-06-16; First posted 2017-07-05 (Actual); Results first posted 2019-10-31 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Rotavirus Infection; Rotavirus Vaccines
Keywords: Immunogenicity; lyophilized formulation; United States; Reactogenicity; Safety; Porcine circovirus -free; Human rotavirus vaccine; liquid formulation; Healthy infants
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine; PEDIARIX; Tetanus Toxoid; Hepatitis B Vaccines; Poliovirus Vaccine, Inactivated; Hiberix; 13-valent pneumococcal vaccine; CRM197 (non-toxic variant of diphtheria toxin)

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HRV PCV-free Liq Group (Experimental): Healthy female or male subjects, between and including 6 and 12 weeks (42-90 days) of age at the time of the first study vaccination who received two doses of oral live-attenuated human rotavirus (HRV) vaccine in PCV-free liquid formulation, according to a 0, 2-month schedule, co-administered with one dose of each Pediarix, Hiberix and Prevnar-13 at three timepoints (day 1, month 2 and month 4). PCV-free implies no detection of PCV-1 and PCV-2 according to the limit of detection of the tests used.
  Interventions: Biological: Rotarix; Biological: Pediarix; Biological: Hiberix; Biological: Prevenar 13
- HRV Lyo Group (Active Comparator): Healthy female or male subjects, between and including 6 and 12 weeks (42-90 days) of age at the time of the first study vaccination who received two doses of oral live-attenuated human rotavirus (HRV) vaccine in lyophilized formulation, according to a 0, 2-month schedule, co-administered with one dose of each Pediarix, Hiberix and Prevnar-13 at three timepoints (day 1, month 2 and month 4).
  Interventions: Biological: Rotarix; Biological: Pediarix; Biological: Hiberix; Biological: Prevenar 13

INTERVENTIONS:
Biological: Rotarix — Two doses administered orally according to a 0, 2 month schedule as per the immunization schedule for HRV vaccine administration in the US.
  Other Names: GSK Biologicals' PCV-free liquid formulation of oral live attenuated HRV vaccine.; GSK Biologicals' lyophilized formulation of oral live attenuated HRV vaccine.
Biological: Pediarix — Three doses administered intramuscularly according to a 0, 2, 4 month schedule.
  Other Names: GSK Biologicals' Diphtheria and tetanus toxoids and acellular pertussis adsorbed; hepatitis B (recombinant) and inactivated poliovirus vaccine.
Biological: Hiberix — Three doses administered intramuscularly according to a 0, 2, 4 month schedule.
  Other Names: GSK Biologicals' Haemophilus b conjugate vaccine (tetanus toxoid conjugate)
Biological: Prevenar 13 — Three doses administered intramuscularly according to a 0, 2, 4 month schedule.
  Other Names: Pfizer's Pneumococcal 13-valent conjugate vaccine (diphtheria CRM197 Protein)

SUMMARY:
The purpose of this study is to assess if there is any immune interference between the Porcine circovirus free (PCV-free) liquid Human rotavirus (HRV) vaccine and routine infant vaccinations currently in use in the US, namely Pediarix®, Hiberix® and Prevenar 13® as compared to the currently licensed lyophilized formulation of the HRV vaccine when co-administered with the same routine vaccinations in healthy infants 6-12 weeks of age

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/[LAR(s)] who, in the opinion of the investigator can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first study vaccination.
* Written or witnessed/thumb printed informed consent obtained from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before the first dose of study vaccines (Day-29 to Day 1), or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone (≥0.5 mg/kg/day, or equivalent). Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before the first dose of vaccine administration and ending at Visit 4, with the exception of the inactivated influenza vaccine, which is allowed at any time during the study, if administered at a site which is different from the sites used to administer the co-administered vaccines.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Uncorrected congenital malformation of the gastrointestinal tract that would predispose for Intussusception (IS).
* History of IS.
* Very prematurely born infants (born ≤28 weeks of gestation).
* Family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Major congenital defects or serious chronic illness.
* Previous vaccination against Haemophilus type b (Hib), diphtheria, tetanus, pertussis, pneumococcus, RV and/or poliovirus.
* Previous confirmed occurrence of RV GE, Hib, diphtheria, tetanus, pertussis, pneumococcus, hepatitis B and/or polio disease.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* GE within 7 days preceding the study vaccine administration.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Hypersensitivity to latex.
* History of any neurological disorders or seizures.
* History of Severe combined immunodeficiency (SCID).
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥38.0°C/100.4°F. The preferred location for measuring temperature in this study will be the oral cavity, the axilla and the rectum.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1280 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (43):
- United States (43):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Boone, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Grove City, Ohio
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Kaysville, Utah
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 48 centers in the United States (US).
Pre-assignment Details: Out of 1280 subjects enrolled in the study, 7 subjects did not receive any study treatment and 1 subject was eliminated from all analyses as there was a deviation in informed consent.
  1272 subjects were vaccinated and included in the Exposed Set, 1148 subjects completed the study.
Groups:
- HRV Porcine Circovirus (PCV)-Free Liquid Group: Healthy female or male subjects, between and including 6 and 12 weeks (42-90 days) of age at the time of the first study vaccination who received two doses of oral live-attenuated human rotavirus (HRV) vaccine in PCV-free liquid formulation, according to a 0, 2-month schedule, co-administered with one dose of each Pediarix, Hiberix and Prevnar-13 at three timepoints (day 1, month 2 and month 4). PCV-free implies no detection of PCV-1 and PCV-2 according to the limit of detection of the tests used.
- HRV Lyophilized Group: Healthy female or male subjects, between and including 6 and 12 weeks (42-90 days) of age at the time of the first study vaccination who received two doses of oral live-attenuated human rotavirus (HRV) vaccine in lyophilized formulation, according to a 0, 2-month schedule, co-administered with one dose of each Pediarix, Hiberix and Prevnar-13 at three timepoints (day 1, month 2 and month 4).
Period: Overall Study
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Started | 632 | 640
Completed | 574 | 574
Not Completed | 58 | 66
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 21 | 29
Not completed — Protocol Violation | 0 | 1
Not completed — CONSENT WITHDRAWAL, NOT DUE TO AN AE | 11 | 13
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 7 | 10
Not completed — NOT WILLING TO PARTICIPATE THIS VISIT | 10 | 5
Not completed — NOT WILLING / NOT ABLE TO BE CONTACTED | 1 | 2
Not completed — OTHER, NOT SPECIFIED | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group | Total
Number analyzed (Participants) | 632 | 640 | 1272
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.7 (1.1) | 8.7 (1.1) | 8.7 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 309 | 617
  Male | 324 | 331 | 655
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 8 | 7 | 15
  Asian | 20 | 22 | 42
  Black Or African American | 74 | 78 | 152
  Native Hawaiian Or Other Pacific Islander | 2 | 2 | 4
  White | 468 | 471 | 939
  Other, not specified | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects With Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations Above or Equal to Cut-off Value.
Description: Immunogenicity was assessed using Enzyme Linked Immunosorbent Assay (ELISA) in terms of seroprotection rates against diphtheria toxoid. A seroprotected subject is a subject whose antibody concentration is greater than or equal to (≥) the level defining clinical protection. The following seroprotection thresholds were applicable:anti-D antibody concentrations ≥ 0.1 International Units/milliliter (IU/mL), anti-T antibody concentrations ≥ 0.1 IU/mL.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: Analysis was performed on the Per protocol set (PPS) for immunogenicity which included all vaccinated subjects for whom immunogenicity data were available, who complied with the procedures and intervals defined in the protocol and for whom assay results were available for antibodies against at least one routine infant vaccine antigen component.
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 486 | 495
Participants
  Anti-D: number analyzed (Participants) | 478 | 486
  Anti-D | 478 | 486
  Anti-T | 486 | 495
Statistical Analysis 1: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of group difference in percentage of subjects with seroprotective concentrations (≥ 0.1 IU/mL) of anti-D antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided asymptotic standardized 95% Confidence Interval (CI) for the difference in seroprotective concentration (HRV PCV-free Liquid group minus HRV Lyophilized group) for each of anti-D antibodies should be ≥-10%; Difference in anti-D concentration = -0.00, 95% CI 2-sided [-0.80 to 0.79]
Statistical Analysis 2: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of group difference in percentage of subjects with seroprotective concentrations (≥ 0.1 IU/mL) of anti-T antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided asymptotic standardized 95% Confidence Interval (CI) for the difference in seroprotective concentration (HRV PCV-free Liquid group minus HRV Lyophilized group) for each of anti-T antibodies should be ≥-10%; Difference in anti-T concentration = -0.00, 95% CI 2-sided [-0.79 to 0.77]

2. Primary Outcome: Number of Seroprotected Subjects With Anti-hepatitis B (Anti-HBs) Antibody Concentrations Above or Equal to Cut-off Value.
Description: Immunogenicity was assessed using ChemiLuminescence ImmunoAssay (CLIA) in terms of seroprotection rates against Hepatitis B. A seroprotected subject is a subject whose antibody concentration is ≥ the level defining clinical protection. The following seroprotection thresholds were applicable:anti-HB antibody concentrations ≥ 10 milli International Units/milliliter (mIU/mL).
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: Analysis was performed on the PPS for immunogenicity which included all vaccinated subjects for whom immunogenicity data were available, who complied with the procedures and intervals defined in the protocol and for whom assay results were available for antibodies against at least one routine infant vaccine antigen component.
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 460 | 471
Participants | 457 | 471
Statistical Analysis 1: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of group difference in percentage of subjects with seroprotective concentrations (≥ 10 mIU/mL) of anti-HB antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided asymptotic standardized 95% CI for the difference in seroprotective concentration (HRV PCV-free Liquid group minus HRV Lyophilized group) for each of anti-HB antibodies should be ≥-10%; Difference in anti-HB concentration = -0.65, 95% CI 2-sided [-1.90 to 0.16]

3. Primary Outcome: Number of Seroprotected Subjects With Anti-polio Virus Types 1, 2 and 3 Antibody Titers Above or Equal to Cut-off Value.
Description: Immunogenicity was assessed using virus micro-neutralization test in terms of seroprotection rates against polio virus types 1, 2 and 3. A seroprotected subject is a subject whose antibody concentration is ≥ the level defining clinical protection. The following seroprotection thresholds were applicable:anti-polio virus types 1, 2 and 3 types antibody titers ≥ 8 Estimated Dose 50% (ED50).
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 477 | 487
Participants
  Anti-Polio 1 | 477 | 486
  Anti-Polio 2: number analyzed (Participants) | 464 | 479
  Anti-Polio 2 | 463 | 478
  Anti-Polio 3: number analyzed (Participants) | 439 | 454
  Anti-Polio 3 | 439 | 454
Statistical Analysis 1: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of group difference in percentage of subjects with seroprotective titers (≥ 8 ED50) of anti-poliovirus type 1 antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided asymptotic standardized 95% CI for the difference in seroprotective concentration (HRV PCV-free Liquid group minus HRV Lyophilized group) for each of anti-poliovirus type 1 antibodies should be ≥-5%; Difference in anti-polio 1 concentration = 0.21, 95% CI 2-sided [-0.60 to 1.15]
Statistical Analysis 2: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of group difference in percentage of subjects with seroprotective titers (≥ 8 ED50) of anti-poliovirus type 2 antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided asymptotic standardized 95% CI for the difference in seroprotective concentration (HRV PCV-free Liquid group minus HRV Lyophilized group) for each of anti-poliovirus type 2 antibodies should be ≥-5%; Difference in anti-polio 2 concentration = -0.01, 95% CI 2-sided [-1.02 to 0.98]
Statistical Analysis 3: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of group difference in percentage of subjects with seroprotective titers (≥ 8 ED50) of anti-poliovirus type 3 antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided asymptotic standardized 95% CI for the difference in seroprotective concentration (HRV PCV-free Liquid group minus HRV Lyophilized group) for each of anti-poliovirus type 3 antibodies should be ≥-5%; Difference in anti-polio 3 concentration = -0.00, 95% CI 2-sided [-0.87 to 0.84]

4. Primary Outcome: Immunogenicity in Terms of Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations.
Description: Antibody concentrations against PT, FHA and PRN were determined and expressed as Geometric Mean Concentrations (GMCs).The GMC calculations were performed by taking the anti-log of the mean of the log concentration transformations.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 486 | 495
IU/mL
  Anti-PT | 51 [47.8 to 54.5] | 54.2 [51.3 to 57.4]
  Anti-FHA | 107.3 [101.4 to 113.5] | 107.7 [101.6 to 114.1]
  Anti-PRN | 55 [50.1 to 60.4] | 56.6 [51.9 to 61.7]
Statistical Analysis 1: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for anti-PT antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for each of anti-PT antibodies should be ≥ 0.67; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 0.94, 95% CI 2-sided [0.86 to 1.03]
Statistical Analysis 2: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for anti-FHA antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for each of anti-FHA antibodies should be ≥ 0.67; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.00, 95% CI 2-sided [0.92 to 1.08]
Statistical Analysis 3: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for anti-PRN antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for each of anti-PRN antibodies should be ≥ 0.67; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 0.97, 95% CI 2-sided [0.86 to 1.10]

5. Primary Outcome: Immunogenicity in Terms of Anti-pneumococcal Serotypes (Anti-PnPS) Antibody Concentrations.
Description: Antibody concentrations against pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) were determined and expressed as GMCs in micrograms per milliliter (µg/mL).The GMC calculations were performed by taking the anti-log of the mean of the log concentration transformations.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 448 | 466
µg/mL
  Anti-PnPS 1 | 1.95 [1.81 to 2.10] | 1.89 [1.76 to 2.03]
  Anti-PnPS 3 | 0.53 [0.49 to 0.57] | 0.53 [0.49 to 0.57]
  Anti-PnPS 4 | 1.24 [1.16 to 1.34] | 1.25 [1.18 to 1.34]
  Anti-PnPS 5: number analyzed (Participants) | 441 | 459
  Anti-PnPS 5 | 1.28 [1.17 to 1.39] | 1.22 [1.13 to 1.31]
  Anti-PnPS 6A | 2.84 [2.64 to 3.05] | 2.8 [2.61 to 3.00]
  Anti-PnPS 6B: number analyzed (Participants) | 448 | 465
  Anti-PnPS 6B | 1.93 [1.72 to 2.15] | 2 [1.80 to 2.22]
  Anti-PnPS 7F | 3.01 [2.83 to 3.21] | 3.04 [2.86 to 3.22]
  Anti-PnPS 9V: number analyzed (Participants) | 447 | 466
  Anti-PnPS 9V | 1.68 [1.56 to 1.81] | 1.63 [1.52 to 1.75]
  Anti-PnPS 14 | 6.27 [5.74 to 6.84] | 6.26 [5.75 to 6.82]
  Anti-PnPS 18C | 1.81 [1.68 to 1.95] | 1.76 [1.64 to 1.89]
  Anti-PnPS 19A | 1.87 [1.73 to 2.02] | 1.8 [1.68 to 1.93]
  Anti-PnPS 19F | 2.94 [2.76 to 3.12] | 2.85 [2.69 to 3.03]
  Anti-PnPS 23F: number analyzed (Participants) | 448 | 462
  Anti-PnPS 23F | 1.14 [1.04 to 1.24] | 1.16 [1.07 to 1.26]
Statistical Analysis 1: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 1; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 1 should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.03, 95% CI 2-sided [0.93 to 1.14]
Statistical Analysis 2: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 3; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 3 should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.00, 95% CI 2-sided [0.91 to 1.11]
Statistical Analysis 3: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 4; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 4 should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 0.99, 95% CI 2-sided [0.90 to 1.09]
Statistical Analysis 4: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 5; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 5 should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.05, 95% CI 2-sided [0.94 to 1.17]
Statistical Analysis 5: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 6A; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 6A should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.01, 95% CI 2-sided [0.92 to 1.12]
Statistical Analysis 6: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 6B; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 6B should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 0.96, 95% CI 2-sided [0.83 to 1.12]
Statistical Analysis 7: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 7F; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 7F should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 0.99, 95% CI 2-sided [0.91 to 1.08]
Statistical Analysis 8: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 9V; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 9V should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.03, 95% CI 2-sided [0.93 to 1.14]
Statistical Analysis 9: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 14; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 14 should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.00, 95% CI 2-sided [0.89 to 1.13]
Statistical Analysis 10: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 18C; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 18C should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.03, 95% CI 2-sided [0.92 to 1.14]
Statistical Analysis 11: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 19A; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 19A should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.04, 95% CI 2-sided [0.93 to 1.15]
Statistical Analysis 12: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 19F; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 19F should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 1.03, 95% CI 2-sided [0.95 to 1.12]
Statistical Analysis 13: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of GMC ratios for Streptococcus pneumoniae (S. pneumoniae) serotype 23F; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% CI on GMC ratios (HRV PCV-free Liquid group over HRV Lyophilized group) for S. pneumoniae serotype 23F should be ≥ 0.5; ANOVA; ANOVA model that included the vaccine group as fixed effect; GMC ratio = 0.98, 95% CI 2-sided [0.87 to 1.10]

6. Primary Outcome: Number of Seroprotected Subjects With Anti-polyribosyl Ribitol Phosphate (Anti-PRP) Antibody Concentrations Above or Equal to Cut-off Value of 0.15 µg/mL.
Description: Immunogenicity was assessed in terms of seroprotection rates against PRP antibodies. A seroprotected subject is a subject whose antibody concentration is ≥ the level defining clinical protection. The following seroprotection thresholds were applicable:anti-PRP antibody concentrations ≥ 0.15 µg/mL.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 485 | 492
Participants | 473 | 479
Statistical Analysis 1: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of group difference in percentage of subjects with concentrations (≥ 0.15 µg/mL) of anti-PRP antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided asymptotic standardized 95% CI for the difference in seroprotective concentrations (HRV PCV-free Liquid group minus HRV Lyophilized group) for each of anti-PRP antibodies should be ≥-5%; Difference in anti-PRP concentration = 0.17, 95% CI 2-sided [-1.94 to 2.28]

7. Primary Outcome: Number of Seroprotected Subjects With Anti-polyribosyl Ribitol Phosphate (Anti-PRP) Antibody Concentrations Above or Equal to Cut-off Value of 1.0 µg/mL.
Description: Immunogenicity was assessed in terms of seroprotection rates against PRP antibodies. A seroprotected subject is a subject whose antibody concentration is ≥ the level defining clinical protection. The following seroprotection thresholds were applicable:anti-PRP antibody concentrations ≥ 1.0 µg/mL.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 485 | 492
Participants | 394 | 404
Statistical Analysis 1: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; Non-inferiority of the immune responses to 3 doses of Pediarix, Hiberix and Prevenar 13 when co-administered with 2 doses of the PCV-free liquid HRV vaccine, as compared to when co-administered with lyophilized HRV vaccine in terms of group difference in percentage of subjects with concentrations (≥ 1.0 µg/mL) of anti-PRP antibodies; Test type: Non-Inferiority — Lower limit (LL) of the two-sided asymptotic standardized 95% CI for the difference in seroprotective concentrations (HRV PCV-free Liquid group minus HRV Lyophilized group) for each of anti-PRP antibodies should be ≥-10%; Difference in anti-PRP concentration = -0.88, 95% CI 2-sided [-5.75 to 3.99]

8. Primary Outcome: Number of Subjects With Seroresponse to Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibodies.
Description: Seroresponse is defined as the percentage of subjects showing an antibody concentration above a threshold that leads to 95% seroresponse in the HRV lyophilized Group. The cut-offs used were as follows: anti-PT (18.566 IU/mL), anti-FHA (35.711 IU/mL) and anti-PRN (11.034 IU/mL).
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 486 | 495
Participants
  Anti-PT | 440 | 470
  Anti-FHA | 466 | 470
  Anti-PRN | 455 | 470
Statistical Analysis 1: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; To rule out 10% decrease in seroresponse to PT antigen in subjects who received Pediarix co-administered with PCV-free-Liquid-HRV vaccine compared to subjects who received Pediarix co-administered with currently licensed lyophilized HRV vaccine where seroresponse was defined as percentage of subjects who showed a concentration above a threshold that led to 95% seroresponse in HRV lyophilized group; Test type: Other — p-value on the difference in seroresponse (HRV PCV-free Liquid group minus HRV Lyophilized group) between groups should be <=0.025 for PT antigen; p < .0001, t-test, 1 sided; p-value was computed by integrating on p-values of 1 sided test with alpha=0.025 & the posterior probability of the cut-off in HRV Lyophilized group
Statistical Analysis 2: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; To rule out 10% decrease in seroresponse to FHA antigen in subjects who received Pediarix co-administered with PCV-free-Liquid-HRV vaccine compared to subjects who received Pediarix co-administered with currently licensed lyophilized HRV vaccine where seroresponse was defined as percentage of subjects who showed a concentration above a threshold that led to 95% seroresponse in HRV lyophilized group; Test type: Other — p-value on the difference in seroresponse (HRV PCV-free Liquid group minus HRV Lyophilized group) between groups should be <=0.025 for FHA antigen; p < .0001, t-test, 1 sided; [statistical method as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: HRV Porcine Circovirus (PCV)-Free Liquid Group vs HRV Lyophilized Group; To rule out 10% decrease in seroresponse to PRN antigen in subjects who received Pediarix co-administered with PCV-free-Liquid-HRV vaccine compared to subjects who received Pediarix co-administered with currently licensed lyophilized HRV vaccine where seroresponse was defined as percentage of subjects who showed a concentration above a threshold that led to 95% seroresponse in HRV lyophilized group; Test type: Other — p-value on the difference in seroresponse (HRV PCV-free Liquid group minus HRV Lyophilized group) between groups should be <=0.025 for PRN antigen; p < .0001, t-test, 1 sided; [statistical method as in outcome 8, analysis 1]

9. Secondary Outcome: Number of Seropositive Subjects With Anti-Rota Virus Immunoglobulin A (Anti-RV IgA) Antibody Concentrations Above or Equal to Cut-off Value of 20 Units/Milliliter (U/mL).
Description: Immunogenicity was assessed in terms of seropositivity against Rota virus IgA antibodies. The cut off used was ≥ 20 U/mL.
Time Frame: At Month 5 (Three months after Dose 2 of HRV vaccine)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 417 | 426
Participants | 318 | 336

10. Secondary Outcome: Number of Seropositive Subjects With Anti-RV IgA Antibody Concentrations Above or Equal to Cut-off Value of 90 U/mL.
Description: Immunogenicity was assessed in terms of seropositivity against Rota virus IgA antibodies. The cut off used was ≥ 90 U/mL.
Time Frame: At Month 5 (Three months after Dose 2 of HRV vaccine)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 417 | 426
Participants | 219 | 238

11. Secondary Outcome: Number of Seropositive Subjects With Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations Above or Equal to Cut-off Value.
Description: Immunogenicity was assessed using ELISA technique in terms of seropositivity against PT, FHA and PRN antibodies. The cut-offs for antibodies were the Lower Limit Of Quantification (LLOQ) of the assays which were ≥ 2.693 IU/mL (anti-PT), ≥ 2.046 IU/mL (anti-FHA) and ≥ 2.187 IU/mL (anti-PRN).
  The Limit of Quantification is the lowest analyte concentration that can be quantitatively detected with a stated accuracy and precision, and LLOQ is the lowest standard curve point obtained by extrapolation, that can still be used for quantification.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 486 | 495
Participants
  Anti-PT | 485 | 495
  Anti-FHA | 486 | 495
  Anti-PRN | 486 | 495

12. Secondary Outcome: Number of Seropositive Subjects With Anti-PnPS Antibody Concentrations Above or Equal to Cut-off Value.
Description: Immunogenicity was assessed using ELISA technique in terms of seropositivity against Pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) antibodies. The cut-off used was ≥ 0.35 µg/mL.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 448 | 466
Participants
  Anti-PnPS 1 | 442 | 463
  Anti-PnPS 3 | 317 | 322
  Anti-PnPS 4 | 434 | 453
  Anti-PnPS 5: number analyzed (Participants) | 441 | 459
  Anti-PnPS 5 | 409 | 424
  Anti-PnPS 6A | 441 | 461
  Anti-PnPS 6B: number analyzed (Participants) | 448 | 465
  Anti-PnPS 6B | 407 | 434
  Anti-PnPS 7F | 448 | 466
  Anti-PnPS 9V: number analyzed (Participants) | 447 | 466
  Anti-PnPS 9V | 431 | 454
  Anti-PnPS 14 | 441 | 454
  Anti-PnPS 18C | 436 | 451
  Anti-PnPS 19A | 438 | 458
  Anti-PnPS 19F | 448 | 465
  Anti-PnPS 23F: number analyzed (Participants) | 448 | 462
  Anti-PnPS 23F | 409 | 425

13. Secondary Outcome: Immunogenicity in Terms of Anti-D and Anti-T Antibody Concentrations.
Description: Antibody concentrations against diphtheria and tetanus were determined and expressed as GMCs. The GMC calculations were performed by taking the anti-log of the mean of the log concentration transformations.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 486 | 495
IU/mL
  Anti-D: number analyzed (Participants) | 478 | 486
  Anti-D | 1.85 [1.72 to 1.98] | 1.88 [1.75 to 2.02]
  Anti-T | 1.88 [1.75 to 2.02] | 1.86 [1.74 to 1.99]

14. Secondary Outcome: Immunogenicity in Terms of Anti-PRP Antibody Concentrations.
Description: Antibody concentrations against PRP were determined and expressed as GMCs. The GMC calculations were performed by taking the anti-log of the mean of the log concentration transformations.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 485 | 492
µg/mL | 4.41 [3.82 to 5.09] | 4.28 [3.71 to 4.94]

15. Secondary Outcome: Immunogenicity in Terms of Anti-HBs Antibody Concentrations.
Description: Antibody concentrations against Hepatitis B were determined and expressed as GMCs. The GMC calculations were performed by taking the anti-log of the mean of the log concentration transformations.
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 460 | 471
mIU/mL | 2031.3 [1834.6 to 2249.0] | 2168.9 [1977.5 to 2378.9]

16. Secondary Outcome: Immunogenicity in Terms of Anti-poliovirus Types 1, 2 and 3 Antibody Titers.
Description: Antibody concentrations against Poliovirus types 1, 2 and 3 were determined and expressed as Geometric Mean Titers (GMTs).
Time Frame: At Month 5 (One month after Dose 3 of co-administered vaccines)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 477 | 487
Titers
  Anti-Polio 1 | 747.2 [673.5 to 828.8] | 728.2 [656.3 to 808.0]
  Anti-Polio 2: number analyzed (Participants) | 464 | 479
  Anti-Polio 2 | 659.6 [587.9 to 740.0] | 699.3 [627.7 to 779.0]
  Anti-Polio 3: number analyzed (Participants) | 439 | 454
  Anti-Polio 3 | 1228.7 [1100.3 to 1372.1] | 1291.6 [1159.1 to 1439.3]

17. Secondary Outcome: Number of Subjects With Any Solicited General Adverse Events (AEs).
Description: Assessed solicited general AEs were cough/runny nose; diarrhoea; fever measured by 3 routes which were oral, axillary and rectal, defined as temperature ≥ 38.0 degrees Celsius (°C); irritability; loss of appetite and vomiting. Any = any solicited general AE irrespective of its intensity grade and relationship to vaccination
Time Frame: During the 8-day (Days 1-8) follow-up period after each HRV vaccination.
Population: Analysis was performed on the Exposed set (ES). The ES included all subjects with at least one study vaccine administration documented. A safety analysis based on the ES included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 632 | 640
Participants
  Cough / Runny Nose (Dose 1), Any | 172 | 180
  Cough / Runny Nose (Dose 2), Any: number analyzed (Participants) | 607 | 609
  Cough / Runny Nose (Dose 2), Any | 224 | 222
  Cough / Runny Nose (Across doses), Any | 305 | 313
  Diarrhea (Dose 1), Any | 39 | 36
  Diarrhea (Dose 2), Any: number analyzed (Participants) | 607 | 609
  Diarrhea (Dose 2), Any | 34 | 26
  Diarrhea (Across doses), Any | 69 | 55
  Fever (Dose 1), ≥ 38.0°C | 36 | 32
  Fever (Dose 2), ≥ 38.0°C: number analyzed (Participants) | 607 | 609
  Fever (Dose 2), ≥ 38.0°C | 64 | 75
  Fever (Across doses), ≥ 38.0°C | 89 | 95
  Irritability / Fussiness (Dose 1), Any | 448 | 458
  Irritability / Fussiness (Dose 2), Any: number analyzed (Participants) | 607 | 609
  Irritability / Fussiness (Dose 2), Any | 440 | 427
  Irritability / Fussiness (Across doses), Any | 523 | 522
  Loss of appetite (Dose 1), Any | 204 | 214
  Loss of appetite (Dose 2), Any: number analyzed (Participants) | 607 | 609
  Loss of appetite (Dose 2), Any | 179 | 178
  Loss of appetite (Across doses), Any | 292 | 293
  Vomiting (Dose 1), Any | 110 | 105
  Vomiting (Dose 2), Any: number analyzed (Participants) | 607 | 609
  Vomiting (Dose 2), Any | 83 | 78
  Vomiting (Across doses), Any | 147 | 148

18. Secondary Outcome: Number of Subjects With Any Unsolicited AEs.
Description: Unsolicited AEs assessed include any AE reported in addition to those solicited during the clinical study. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms were reported as an unsolicited AE. Any= Any unsolicited AE irrespective of its intensity grade and relationship to vaccination.
Time Frame: During the 31-day (Days 1-31) follow-up period after each HRV vaccination.
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 632 | 640
Participants | 294 | 327

19. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs).
Description: SAEs assessed include any untoward medical occurrence that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization or resulted in disability/incapacity.
Time Frame: During the entire study period (Day 1 to Month 10)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
Number analyzed (Participants) | 632 | 640
Participants | 20 | 19

ADVERSE EVENTS:
Time Frame: Solicited AEs: During the 8-day (Day 1 to Day 8) follow-up period after each HRV vaccination. Unsolicited AEs: During the 31-day (Day 1 to Day 31) follow-up period after each HRV vaccination. SAEs: Throughout the study period (Day 1 to Month 10).
Arm/Group | HRV Porcine Circovirus (PCV)-Free Liquid Group | HRV Lyophilized Group
All-Cause Mortality (participants affected / at risk) | 1/632 | 0/640
Serious Adverse Events (participants affected / at risk) | 20/632 | 19/640
Other Adverse Events (participants affected / at risk) | 571/632 | 589/640
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HRV Porcine Circovirus (PCV)-Free Liquid Group (N=632) | HRV Lyophilized Group (N=640)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 2 (2)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0)
Botulism (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 5 (5) | 4 (4)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid intake reduced (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (2)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Laryngomalacia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3 (3) | 4 (4)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1)
Rhinovirus infection (Infections and infestations) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HRV Porcine Circovirus (PCV)-Free Liquid Group (N=632) | HRV Lyophilized Group (N=640)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital musculoskeletal anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital torticollis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Macrocephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Plagiocephaly (Congenital, familial and genetic disorders) | 7 (7) | 9 (9)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 8 (9) | 2 (2)
Otorrhoea (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 5 (5) | 1 (1)
Eye discharge (Eye disorders) | 6 (8) | 6 (6)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Eyelid irritation (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (10) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 126 (185) | 113 (164)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 12 (17) | 13 (15)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 (13) | 13 (13)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infantile vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 2 (2)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pylorospasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 12 (12) | 10 (11)
Vomiting (Gastrointestinal disorders) | 155 (208) | 156 (197)
Crying (General disorders) | 3 (3) | 0 (0)
Discomfort (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 2 (2)
Injection site discomfort (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 1 (1)
Injection site inflammation (General disorders) | 0 (0) | 1 (1)
Injection site mass (General disorders) | 1 (1) | 1 (1)
Injection site nodule (General disorders) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 13 (16) | 9 (11)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Nodule (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 102 (116) | 116 (133)
Swelling (General disorders) | 2 (2) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 1 (1) | 2 (2)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 16 (16) | 16 (16)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 5 (5)
Candida nappy rash (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 14 (14) | 11 (11)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 6 (6) | 4 (4)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Ear infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 2 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 4 (4)
Gastroenteritis (Infections and infestations) | 7 (7) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 9 (9)
Laryngitis (Infections and infestations) | 0 (0) | 2 (2)
Laryngotracheitis obstructive (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 10 (10)
Neonatal candida infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 6 (6) | 7 (8)
Otitis media (Infections and infestations) | 26 (28) | 23 (26)
Otitis media acute (Infections and infestations) | 14 (14) | 23 (25)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 10 (10)
Respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 4 (5)
Rhinovirus infection (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3)
Skin bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Skin candida (Infections and infestations) | 3 (3) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Subglottic laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 63 (72) | 69 (77)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urogenital infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 8 (9) | 8 (8)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 1 (1)
Viral test positive (Investigations) | 1 (1) | 0 (0)
Breast milk substitute intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cow's milk intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 293 (384) | 293 (392)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Milk soy protein intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Torticollis (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Drooling (Nervous system disorders) | 1 (1) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1)
Poor quality sleep (Nervous system disorders) | 3 (3) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 7 (7) | 5 (5)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 523 (896) | 522 (896)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral discharge (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital labial adhesions (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Penile adhesion (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Testicular retraction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 320 (423) | 330 (446)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 28 (31) | 40 (47)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 21 (21)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Acne infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (10)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 14 (15) | 17 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (3)
Eczema infantile (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 12 (15)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT03207750/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT03207750/SAP_001.pdf